CLINICAL TRIAL: NCT05366582
Title: A Comparison of the Videolaryngoscope and Macintosh Laryngoscope for NIM-EMG Endotracheal Tube Placement: Prospective, Double Blind, Randomized Study
Brief Title: Neural Integrity Monitor Electromyogram (NIM-EMG) Endotracheal Tube Intubation With Video Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, İsmail SÜMER, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Ismail02
Record Dates: First submitted 2022-04-29; First posted 2022-05-09 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Intubation; Difficult or Failed; Airway Complication of Anesthesia; Pain, Postoperative; Anesthesia Intubation Complication
Keywords: Videolaryngoscopy; NIM-EMG intubation tube; thyroidectomy; airway management
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Anesthesia approach appropriate to the group of the randomized patient before the operation will be selected. The chosen intubation method will be performed by the 1st anesthetist. The patient, the surgeon and the second anesthetist who will follow up intraoperatively and postoperatively will not know the chosen method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Macintosh Laryngoscope (ML) (Active Comparator): Macintosh laryngoscope is used for intubation after anesthesia induction
  Interventions: Device: Macintosh Laryngoscope
- Group Video Laryngoscope (VL) (Active Comparator): Video laryngoscope is used for intubation after anesthesia induction
  Interventions: Device: Video Laryngoscope

INTERVENTIONS:
Device: Macintosh Laryngoscope — After the induction, laryngoscopy will be performed with a Macintosh laryngoscope after 2 minutes of manual ventilation after muscle relaxant by an anesthesiologist with at least 4 years of experience. Patients will be intubated with the "Medtronic Xomed Nerve Integrity Monitor Standard Reinforced ElectromyographyEndotracheal Tube" (size 6.0, 7.0 or 8.0). The cuff of the intubation tube will be connected to a manometer and inflated at a pressure of 20-30 mmHg until there is no air leak. Intubation will be confirmed by the appearance of end-tidal carbon dioxide (CO2). Failed intubation will be considered if not achieved within 2 minutes
  Arms: Group Macintosh Laryngoscope (ML)
Device: Video Laryngoscope — After the induction, laryngoscopy will be performed with a Video laryngoscope after 2 minutes of manual ventilation after muscle relaxant by an anesthesiologist with at least 4 years of experience. Patients will be intubated with the "Medtronic Xomed Nerve Integrity Monitor Standard Reinforced ElectromyographyEndotracheal Tube" (size 6.0, 7.0 or 8.0). The cuff of the intubation tube will be connected to a manometer and inflated at a pressure of 20-30 mmHg until there is no air leak. Intubation will be confirmed by the appearance of end-tidal CO2. Failed intubation will be considered if not achieved within 2 minutes
  Arms: Group Video Laryngoscope (VL)

SUMMARY:
Laryngeal nerve monitoring is performed to prevent intraoperative nerve damage in thyroidectomy operations. NIM-EMG intubation tube is used while monitoring the recurrent laryngeal nerve. Care should be taken when placing this tube. Ensure that the electrodes on the tube are in contact with the vocal cords. Both the macintosh laryngoscope and the videolaryngoscope can be used when inserting the NIM-EMG tube. The aim of our study is to compare these two intubation methods.

DETAILED DESCRIPTION:
Anesthesiologists play a key role for the medications used for anesthesia and placement of the endotracheal tube in operations with intraoperative monitoring. While placing the NIM-EMG tube, the size of the endotracheal tube is very important so that the tube can contact the vocal cords.

The placement of the tube may change due to reasons such as movement of the neck during the operation. In addition, endotracheal tube placement may be problematic due to poor vision during direct laryngoscopy. Incorrect placement of the tube may result in equipment inoperability and increase the likelihood of injury to the recurrent laryngeal nerve.

Laryngoscopy is a term for tracheal intubation that provides visualization and evaluation of the larynx with its upper airway structures.

Until recently, direct laryngoscopy was considered the standard technique for endotracheal intubation. Recently, a wide variety of methods have been developed for endotracheal intubation. Video laryngoscopes are similar to direct laryngoscopes but provide laryngeal imaging with a small video chip on their blade. This imaging is superior compared to direct laryngoscopy. The aim of the study was to compare the use of direct laryngoscopy and video laryngoscopy in intubation with the NIM-EMG tube, which is routinely used in operations where the recurrent laryngeal nerve (RLN) may be damaged, in terms of intubation success, intubation time, tracheal intubation comfort, hemodynamic responses, surgical satisfaction, and complications that may develop after anesthesia or surgery.

ELIGIBILITY:
Inclusion Criteria:

* The American Society of Anesthesiologists (ASA) physical status classification system 1-2
* Age 18-65
* Undergoing Elective Thyroid and Parathyroidectomy surgery
* undergoing Intraoperative Recurrent Laryngeal Nerve Monitoring

Exclusion Criteria:

* History of head and neck surgery
* Body mass index less than 19 or greater than 30
* Muscle relaxant allergy
* Lidocaine allergy
* IDS score >5
* Uncontrolled hypertension, bronchial asthma, tracheal pathology
* undergoing emergency surgery
* Cases that cannot give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Number of intubation attempts | during intubation after induction of anesthesia
  The number of intubation attempts between both groups will be recorded. that patients are intubated will be confirmed by the presence of end tidal carbon dioxide.
Difficulty of Laryngoscopy | during intubation after induction of anesthesia
  The Helbo-Hansen scoring system-Steyn Modification will be used to determine the quality of laryngoscopy.
  Helbo-Hensen et al. with Steyn modification includes five criteria; ease of laryngoscopy, degree of coughing, position of vocal cords, jaw relaxation, and limb movement and graded on a 4-point scale.Total score of 5 will considere to be excellent, 6-10 good, 11-15 poor, and 16-20 bad. Total scores will divide into clinically acceptable and not acceptable scores (total score ≤ 10 acceptable, >10 unacceptable).
Difficulty of Intubation | during intubation after induction of anesthesia
  The intubation difficulty scale (IDS) of patients will be used to determine the difficulty of intubation during laryngoscopy, and the Helbo-Hansen scoring system-Steyn Modification will be used to determine the quality of laryngoscopy.
  Intubation Difficulty Scale (IDS) score, which is a function of seven parameters, resulting in a progressive, quantitative determination of intubation complexity.
  intubation difficulty may be defined as a measure of the degree of divergence from a predefined "ideal" intubation, i.e., one performed without effort, on the first attempt, practiced by one operator, using one technique, with full visualization of the laryngeal aperture and vocal cords abducted. Such an intubation is accorded an IDS value of 0. Each variation from this defined "ideal" intubation increases the degree of difficulty, the overall score being the sum of all variations from this definition. Impossible intubation is defined by infinity (IDS =[infinity]).
NIM-EMG tube placement success | during intubation after induction of anesthesia
  After placing the special tube and checking its level and contact, the grounding subdermal needle electrodes will be placed on the shoulder and all of the electrodes will be connected to the main unit. The impedance of the electrodes will be measured and the tube will be fixed after the device confirms that the impedance values are below 4 kiloohm (kΩ).
Intubation time | during intubation after induction of anesthesia
  After anesthesia induction and muscle relaxant, the time will be started when patients who are manually ventilated for 2 minutes are ready for intubation. When successful intubation is proven, the time will be stopped and the duration recorded.

SECONDARY OUTCOMES:
sore throat | up to 24 hours postoperative period
  Sore throat of the patients was evaluated as present or absent at the postoperative 30th minute, 2,6 and 24 hours by the patient.
dysphagia | up to 24 hours postoperative period
  dysphagia of the patients was evaluated as present or absent at the postoperative 30th minute, 2,6 and 24 hours by the patient.
patient satisfaction | up to 24 hours postoperative period
  It will be evaluated by the patient between zero and ten points according to the patient satisfaction scale and the severity of sore throat and hoarseness. The patient satisfaction score is scored over a minimum of 0 points and a maximum of 10 points. A score of 0 means I am not satisfied at all, a score of 10 means very satisfied. A higher score indicates higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Sumer, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)